CLINICAL TRIAL: NCT02943434
Title: Diet-Induced Thermogenesis: A Comparison of Whole and Processed Foods
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Central Washington University (Other)
Responsible Party: Principal Investigator, Nicole Stendell-Hollis, Assistant Professor, Central Washington University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 161020
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Food, Processed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Processed Food (Other): Changes in resting energy expenditure will be measured via indirect calorimetry after consumption of a processed foods meal to determine changes in diet-induced thermogenesis.
  Interventions: Other: Processed food
- Whole Food (Other): Changes in resting energy expenditure will be measured via indirect calorimetry after consumption of a whole foods meal to determine changes in diet-induced thermogenesis.
  Interventions: Other: Processed food

INTERVENTIONS:
Other: Processed food — This is examining the effects of processed foods on diet-induced thermogenesis.

SUMMARY:
This study will examine differences in diet-induced thermogenesis (DIT) between a meal made of processed ingredients and an equivalent, isocaloric meal made of whole ingredients. For the purpose of this study processed foods (PFs) will be considered those that are purchased in a state that is modified from their whole food (WF) counterpart (e.g. shell eggs compared to powdered eggs). Research has shown that less energy is expended to digest processed foods than whole foods, which confers an advantage to processed foods in terms of caloric efficiency, but a disadvantage in terms of energy balance and weight loss. A 2010 study showed that subjects expended approximately 10% less energy to digest sandwiches made of white bread and cheese product compared to sandwiches made of whole grain bread and cheddar cheese. The intent of this study is to enhance those results and improve upon the study design by constructing meals to be more similar in the makeup of individual ingredients, making ingredient processing a more isolated variable. Subjects will be healthy CWU male students with a body mass index of 18.5 - 24.9 kg/m2. Metabolism will be assessed by repeated measurements of resting energy expenditure via indirect calorimetry. Measurements of baseline metabolism will be made; subjects will then be provided one of two meals, both comprised of rice, green beans, and eggs cooked in canola oil and equivalent but differing in processing status (e.g. brown rice and white rice, fresh cooked green beans and canned green beans, etc). Hourly metabolic measurements will be made post-meal for 6 hours. During this time subjects will be asked to minimize non-DIT deviations in metabolism; e.g. those due to physical activity, excitement level, etc. The procedure will be repeated one week later with the other meal so that changes in DIT can be assessed on a subject-by-subject basis. The results of this study will be assessed in the lens of weight loss, specifically dietary choices that affect energy balance. It is possible that consuming a diet that includes more whole foods (versus processed foods) would be beneficial to the attainment of a healthy body weight - either through potential weight loss or weight maintenance.

DETAILED DESCRIPTION:
This study will be a crossover design that will use indirect calorimetry to assess changes in metabolic rates in twelve healthy subjects prescreened for any known metabolic abnormalities. Subjects will be recruited from healthy CWU male students of a normal BMI range that express interest in research study participation. Subjects will be assigned either a meal made of whole ingredients (whole grain brown rice, unrefined canola oil, scrambled eggs from the shell, freshly-steamed green beans) or one made of processed ingredients (white rice, canola oil-based margarine, scrambled eggs from a powdered mix, canned green beans). Subjects will have a basal metabolic rate (BMR) measurement taken before ingesting the meal and DIT will be measured on an hourly basis post meal.

PROCEDURE:

Early Meal Preparation:

Meal preparation will begin the night prior to each testing session by cooking 2 cups of dry rice per the package instructions and chilling it in a shallow stainless steel pan. This rice will be refrigerated overnight and re-heated portion-by-portion for the following morning's meal feeding. Three portions of one cup's worth of fresh green beans will also be washed, trimmed, cut into one-inch pieces, and refrigerated.

Initial Testing:

Two subjects will be assessed per day. Subjects will each report to the lab for a total of two days (approximately 8 hour days) one week apart for a baseline metabolic measurement, a meal feeding, and a series of post-meal metabolic measurements. Measurements will take 30 minutes to complete, including time for calibration to the individual prior to the measurement and time for cleaning and preparing the assessment equipment for the next subject. Subjects will arrive in thirty minute staggered scheduled intervals each morning (see proposed example schedule attached). At least three days prior to initial testing subjects will be provided with a three-day diet intake record to be completed by the subject during the three days prior to initial testing. Instructions on correct completion of the three day diet record will be given to each subject when they are provided with the three day records (please see attached; this diet record has been modified and used with permission from the Colorado Clinical and Translational Sciences Institute-[see attached email]). At this time subjects will be re-briefed on pre-test protocol and provided instructions for setting up and using the heart rate monitors. The three day records will be reviewed with each subject on the day of data collection for completeness and accuracy.

Pre-test protocol:

Protein has the greatest effect on metabolism of all macronutrients, so intake will be limited to no more than the recommended daily allowance of .8 g protein per kg body weight3 the evening prior to testing; all other macronutrient and micronutrient intakes are to be consumed at the discretion of the subject. No intake with caloric content is to be consumed after a point in the evening which is 12 hours prior to testing (approximately 7 PM). Subjects will be asked to abstain from alcohol, marijuana, and caffeine use the night before and the day of testing. Subjects will be asked to refrain from strenuous physical activity for two days before testing and to restrain from all but light physical activity the day before testing. Upon awakening the morning of testing, subjects will activate a MyZone MZ-3 heart rate monitor and consume 500 mL of supplied bottled water. Subjects will report to the lab, expending as little energy as possible (driving instead of walking, taking the elevator instead of stairs, etc).

Resting Phase and BMR:

Upon arriving at the testing site, subjects will be provided a 30 minute period during which they will be briefed again on the procedure, allowed to urinate or defecate if needed, and rest until baseline testing. A ParvoMedics TrueOne 2400 Metabolic Measuring System (MMS) will be used to determine metabolic rates using the dilution method outlined in the manual (see attached). At the beginning of the 30 minute BMR testing period the subject will lie face up on the assessment table and will be allowed to get comfortable before being fitted with the measurement hood. The flow rate of the MMS dilution pump will be calibrated to each subject. During each measurement, the subject will be instructed to lie still with the eyes closed while breathing normally.

Immediate Meal Preparation:

Whole Food Meals Bring one quart of water to boil in a medium pot. Heat 2 Tbsp unrefined canola oil on medium heat in a skillet. Beat 3 large shell eggs together in a cup and add directly to the skillet, cooking and stirring until eggs are fluffy and set (3-5 minutes). During this time, place 1 cup of cut green beans in a metal strainer, set above boiling water, and cover with lid for 3 minutes. Place 1.5 cups of precooked brown rice on a plate and microwave for 1.5 minutes, then allow to stand for 2 minutes to ensure even heating. Add cooked eggs and green beans to plate, and scrape oil over rice with a spatula. Cover plate with a lid and deliver to testing site. Microwave meal for 30 seconds immediately before serving.

Processed Food Meals:

Drain and rinse 1 cup of canned green beans. Heat 2 Tbsp canola-based margarine on medium heat in a skillet. Prepare 3 eggs' worth of powdered egg mix per package instructions and add directly to the skillet, cooking and stirring until eggs are fluffy and set (3-5 minutes). During this time, place 1.5 cups of precooked white rice and the 1 cup of green beans on a plate and microwave for 1.5 minutes, then allow to stand for 2 minutes to ensure even heating. Add cooked eggs to plate, and scrape oil over rice with a spatula. Cover plate with a lid and deliver to testing site. Microwave meal for 30 seconds immediately before serving.

Note: Meal ingredient amounts may change based on the average energy needs of the subjects (e.g. 1 cup of rice instead of 1.5, etc). Both meals will be adjusted so as to keep them isocaloric.

Meal Feeding and Rest:

Subjects will be served one type of meal during the assessment session, and the other meal one week later during the second assessment. Meals will be served immediately after BMR measurements are complete. Subjects will be asked to consume the entire meal and will be provided 30 minutes to do so. Following completion of the meal, subjects will be asked to remain onsite and will be instructed to lie down or sit quietly and rest until the first DIT measurement takes place. During the meal and until the completion of the day's testing, subjects will be permitted to consume only water. A graduated water bottle will be provided to record water intake.

DIT Measurement and Rest:

DIT will be assessed in the same fashion as BMR. The first DIT reading will take place one hour from the beginning of the BMR measurement. Afterwards, subjects will be asked to remain onsite and will be instructed to rest. Subjects may lie down or sit quietly, or engage in a non-physical activity that does not induce psychological stress or excitement. This includes but is not limited to: using the bathroom, reading, completing homework, watching an appropriate movie, talking quietly, etc. DIT measurements will be taken on an hourly basis for six hours or until metabolism returns to base levels. No intake except for water will be permitted until the day's measurements are complete.

Data Analysis:

All subjects will be assigned a study ID number and all data collected will only be identifiable by that study ID number. Only the primary investigators will have access to participant's contact information to assure confidentiality. Summary statistics (mean, standard deviations, ranges, and proportions) will be calculated for baseline demographic characteristics (see attached questionnaire). Three-day diet record information will be entered on ESHA Food Processor Software and quantitative analysis of macronutrient intake performed. Data from the MSM will be transferred on to a Microsoft Excel spreadsheet and repeated measures t-tests performed on metabolic statistics for each subject. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Ages 18 - 25 years
* BMI: 18.5 - 29.9 kg/m2

Exclusion Criteria:

* Diagnosed with cardiovascular disease, cancer, diabetes, thyroid disorder, metabolic disorders, eating disorders, and/or egg allergy

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Changes in resting energy expenditure will be assessed via indirect calorimetry | Resting energy expenditure will be assessed at baseline and post-baseline at hours 1, 2, 3, 4, 5, & 6 for a total of 7 measurements

CONTACTS AND LOCATIONS:
Overall Officials: Nicole R Stendell-Hollis, PhD, Study Chair — Central Washington University

IPD SHARING:
Plan to Share IPD: No